CLINICAL TRIAL: NCT05108935
Title: Providing A Resource: Telemedicine at Needle Exchanges to Reach Under-served Populations - Greensboro
Brief Title: Providing PrEP, Hepatitis C Treatment, and MOUD Through Telemedicine at Greensboro SSP
Acronym: PARTNERUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Center for AIDS Research (CFAR) (Unknown); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00104147_1; 5P30AI064518-17 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-01

CONDITIONS: Opioid Use; Opioid Use Disorder; Risk Reduction; Hiv; Hepatitis C
Keywords: opioid; medication for opioid use disorder; Drug user health hub; syringe services program; syringe exchange; PrEP; HIV prevention; retention in care; Suboxone; Hepatitis C treatment; hepatitis C; Opioid use disorder; feasibility; acceptability
MeSH Terms: conditions — Opioid-Related Disorders; Risk Reduction Behavior; Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — Buprenorphine, Naloxone Drug Combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Pre-Exposure Prophylaxis; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medication and telemedicine follow up (Experimental): Enrolled participants will be prescribed PrEP Mavyret and/or Suboxone. Follow up visits will be conducted by telemedicine. We are testing whether telemedicine is a feasible method for follow up.
  Interventions: Drug: Suboxone; Drug: Truvada; Drug: Mavyret

INTERVENTIONS:
Drug: Suboxone — Enrolled participants will be prescribed PrEP Mavyret and/or Suboxone. Follow up visits will be conducted by telemedicine. We are testing whether telemedicine is a feasible method for follow up.
  Other Names: Buprenorphine Naloxone
Drug: Truvada — Enrolled participants will be prescribed PrEP Mavyret and/or Suboxone. Follow up visits will be conducted by telemedicine. We are testing whether telemedicine is a feasible method for follow up.
  Other Names: Pre-Exposure Prophylaxis (PrEP)
Drug: Mavyret — Enrolled participants will be prescribed PrEP Mavyret and/or Suboxone. Follow up visits will be conducted by telemedicine. We are testing whether telemedicine is a feasible method for follow up.
  Other Names: Hepatitis C treatment

SUMMARY:
The purpose of this study is to provide medication for opioid use disorder (MOUD) with buprenorphine and naloxone, or bup/nx, pre-exposure prophylaxis (PrEP) for HIV prevention, and/or hepatitis C treatment for persons who inject opioids accessing syringe services programs (SSPs), as part of a comprehensive harm reduction program, and assess the acceptability and feasibility of using telemedicine to implement the program.

The initial visit will be conducted in person or remotely via telemedicine given COVID-19 protocols at the SSP site in Greensboro, North Carolina (NC); follow-up visits will be conducted via telemedicine.

DETAILED DESCRIPTION:
The purpose of this study is to provide medication for opioid use disorder (MOUD) with buprenorphine and naloxone, or bup/nx, pre-exposure prophylaxis (PrEP) for HIV prevention and/or hepatitis C treatment for persons who inject opioids accessing syringe services programs (SSPs), as part of a comprehensive harm reduction program, and assess the acceptability and feasibility of using telemedicine to implement the program.

The study objectives are the following:

To assess uptake and persistence to bup/nx, PrEP, and hepatitis C treatment as part of a comprehensive telemedicine-based harm reduction program among people who inject drugs using SSPs.

To assess feasibility and acceptability of implementing a telemedicine-based care harm reduction program among program implementers To assess feasibility and acceptability of participating in a telemedicine-based harm reduction program among users

The study population is people who inject drugs, specifically opioids, and who access services at an SSP in Greensboro, NC. The study team will enroll 30 people who inject drugs accessing the participating SSP. Participants will be enrolled in the study for 6 months. At the end of the study, they will be referred to MOUD and PrEP providers identified in the community.

Data collection

Enrollment visit:

The study coordinator will administer a baseline survey to collect demographics, HIV risk behaviors, and substance use history. Participants will undergo laboratory testing at the SSP to determine eligibility and enrolled participants will be prescribed bup/nx and PrEP free of charge.

Follow up visits:

Follow-up visits will be conducted via telemedicine at the SSP.

Participants on any combination of treatment including MOUD:

For the first month (Month 1), telemedicine visits will be weekly with each to ensure that participants are stable on the appropriate bup/nx dose. Starting at Month 2, the telemedicine visits will take place monthly.

For participants on any combination of treatment NOT including MOUD:

Participants will attend telemedicine follow up visits at month 3 and month 6 to check in and provide labs.

All participants will be asked to complete a questionnaire at Month 3 and Month 6 which include questions on HIV risk and drug use, as well as adherence evaluation. All participants will also be asked to participate in qualitative interviews on their experiences with the program at month 1 and month 6.

By the end of the study, we hope to determine the following:

1. The proportion of persons who demonstrate no or minimal opioid use 1a. Defined as completing Month 3 and Month 6 visits with self-reported opioid use on ≤4 days in the past month and/or 2
2. The proportion of persons who remain HIV negative. 2a.Measured via negative HIV test at Month 3 and Month 6
3. Among participants who undergo hepatitis C treatment, the hepatitis C cure rate
4. Retention or persistence in care 4a. Defined as the proportion who remain on treatment (all or any combination of MOUD, PrEP, and hepatitis C treatment) at Month 3 and Month 6 4b. We will also examine whether participants are more apt to remain on paired/combined therapy compared to individual treatment.
5. Organizational facilitators and barriers to establishing a telehealth program in an SSP 5a. We will iteratively collect programmatic data and document challenges and problem-solving that occurs throughout the implementation period of providing bup/nx, PrEP, and/or hepatitis C treatment. We will identify and describe organizational factors using the framework of the Implementation Research Logic Model.
6. Patient perspectives on telehealth delivery of PrEP, MOUD, and/or hepatitis C treatment via SSP 6a. Analysis of interview data at Month 1 and Month 6 to measure attitudes toward PrEP, MOUD, and hepatitis C treatment in general, and on delivery of treatment via telehealth and at the SSP 6b. Analysis of questionnaire data at baseline, Month 3, and Month 6

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Participant in SSP
* History of self-report injection opioid use in the past 6 months
* Willing to take bup/nx, PrEP, and/or hepatitis C treatment for 6 months
* Not currently taking PrEP
* HIV negative
* Not pregnant
* Either a history of sharing injection or drug preparation equipment or risk of sexual acquisition of HIV* in the past 6 months

  *Individuals are considered at risk of sexual acquisition of HIV if they answer yes to any of the items in the below question: In the last 6 months, have any of the following applied to you?
* Traded sex for money or drugs
* Had a sexual partner who is HIV positive
* Did not consistently use condoms when having sex
* Had a bacterial sexually transmitted infections (like gonorrhea, chlamydia, or syphilis)
* No medical contraindications for these medications such as history of renal failure or bone diseases

Exclusion Criteria:

* Have altered mental status in which participant cannot sign a consent form
* Receive a positive pregnancy test (will be checked at screening visit)
* Receive a positive HIV test at enrollment (will be checked at screening visit)
* Have evidence of renal failure (will be checked at screening visit)
* Have a history of hepatitis B (will be checked at screening visit)
* Becoming incarcerated during the study

Additional considerations:

The following are not exclusion criteria for the study overall, but will affect which treatment(s) they can receive:

* Are currently receiving some form of MOUD (buprenorphine, naltrexone, methadone) - this makes them ineligible for MOUD treatment through the study, but they can still receive PrEP and/or hepatitis C treatment
* Have received treatment for hepatitis C prior to enrollment - this makes them ineligible for hepatitis C treatment through study, but they can still receive PrEP and/or MOUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion who demonstrate no or minimal opioid use. | 3 months
  Defined as self-reported opioid use on ≤4 days in the past month and/or 2 or more consecutive negative urine tests.
Proportion who demonstrate no or minimal opioid use. | 6 months
  Defined as self-reported opioid use on ≤4 days in the past month and/or 2 or more consecutive negative urine tests.
Proportion who remain HIV negative. | 3 months
  Measured via negative HIV test.
Proportion who remain HIV negative. | 6 months
  Measured via negative HIV test.
Among participants who undergo hepatitis C treatment, the hepatitis C cure rate | 6 months
  Measured via negative hepatitis C test.
Persistence in care | 3 months
  Defined as the proportion who remain on treatment.
Persistence in care | 6 months
  Defined as the proportion who remain on treatment.
Ease/difficulty of visiting a SSP to meet with a provider via telemedicine | month 1
  Exploratory method, conducted in the form of individual interviews to document the personal experiences of each participant (qualitative method)
Ease/difficulty of visiting a SSP to meet with a provider via telemedicine | month 6
  Exploratory method, conducted in the form of individual interviews to document the personal experiences of each participant (qualitative method)
Ease/difficulty of accessing the telemedicine video platform | month 1
  Exploratory method, conducted in the form of individual interviews to document the personal experiences of each participant (qualitative method)
Acceptability of medical care via a telemedicine video platform | 6 month
  Exploratory method, conducted in the form of individual interviews to document the personal experiences of each participant (qualitative method)
Participant satisfaction with the program | 1 month
  Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant (qualitative method)
Participant satisfaction with the program | month 6
  Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant over time (qualitative method)
Participant perceived usefulness of the program | month 1
  Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant (qualitative method)
Participant perceived usefulness of the program | month 6
  Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant (qualitative method)
Motivators and barriers affecting program persistence | month 6
  Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant over time (qualitative method)
Motivators and barriers affecting medication adherence and persistence | 6 months
  Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant over time (qualitative method)

CONTACTS AND LOCATIONS:
Overall Officials: Mehri McKellar, MD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Duke Department of Population Health Sciences, Durham, North Carolina
  - NC Survivors Union, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No
We will not share IPD with other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT05108935/ICF_000.pdf